CLINICAL TRIAL: NCT01403584
Title: Adjustment of Non-invasive Positive Pressure Ventilation in Patients With Chronic Hypercapnic Ventilatory Failure Using Automated End-expiratory Pressure (AutoEEP) Algorithm
Brief Title: Adjustment of Mask Pressure, for Bilevel Positive Airways Pressure Therapy, by Automated Algorithm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ResMed (Industry)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 09-4225
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Respiratory Insufficiency; Sleep Disordered Breathing
Keywords: Breathing pattern; Gas exchange; Sleep quality
MeSH Terms: conditions — Respiratory Insufficiency; Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AutoVPAP with addition of AutoEPAP (Experimental): This arm will receive conventional device modified to enable algorithm for automatically applied Expiratory Positive Airway Pressure. Patients randomised to this group will then receive the other treatment the following night.
  Interventions: Device: AutoVPAP with addition of AutoEPAP; Device: AutoVPAP with EPAP manually selected
- AutoVPAP without addition of AutoEPAP (Active Comparator): This arm will receive conventionally applied Expiratory Positive Airway Pressure. Patients randomised to this group will then receive the other treatment the following night.
  Interventions: Device: AutoVPAP with addition of AutoEPAP; Device: AutoVPAP with EPAP manually selected

INTERVENTIONS:
Device: AutoVPAP with addition of AutoEPAP — Implementation of automated algorithm for adjustment of conventional device parameter (EPAP0.
Device: AutoVPAP with EPAP manually selected — Conventionally applied Expiratory Positive Airway Pressure (EPAP)

SUMMARY:
The aim of the study is to test the hypothesis that an automated algorithm for desired mask pressure improves breathing pattern and sleep quality in patients with hypercapnic ventilatory failure. For this purpose, The investigators will study different groups of patients, including those with obstructive and restrictive ventilatory defect, and obstructive sleep apnoea, non-naive to conventional bi-level positive airways pressure therapy.

DETAILED DESCRIPTION:
Persisting ventilatory failure associated with chronic obstructive pulmonary disease (COPD), obesity-hypoventilation-syndrome, sleep apnoea or neuromuscular disease is increasingly managed with domiciliary non-invasive positive pressure ventilation (NIPPV).

Optimal settings of non-invasive ventilation are usually titrated manually and require time and expertise. The development of systems lead to automated analysis and development of algorithms to adjust ventilators. However, there is a paucity of optimal algorithms, particularly the problem of upper airway obstruction. Therefore, the central aim of this study is to develop the automated setting of an end-expiratory positive airway pressure (EPAP), because upper airway obstruction is relatively common in this group of patients. We hypothesise that an automated end-expiratory airway pressure (AutoEEP) adjusting algorithm could overcome these problems and further optimise and adjust ventilator settings. Using non-invasive ventilation in patients with hypercapnic ventilatory failure, awake and asleep, we will measure physiological outcome parameters and apply an AutoEEP algorithm, comparing it against usual care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be patients not naive to noninvasive ventilation, and being so treated for any form of hypercapnic ventilatory failure.
* Previously stabilised on bilevel noninvasive pressure support ventilation.
* Both genders, age <75years.
* Previously shown to have a requirement for an EEP above cm H2O in order to maintain upper airway patency, or those in whom such a raised EEP would be expected, e.g. obese patients.
* Patients also known to have adequate airway patency at an EEP of 4 to 5 cm H2O will be included to ensure specificity of the algorithm.

Exclusion Criteria:

* Acute critical illness (e.g. acute coronary syndrome, stroke)
* Serious anatomical variations of nose, sinuses, pharynx or oesophagus.
* Any condition at risk of oesophageal bleeding (e.g. oesophageal varices, gastric ulcer, etc.)
* Age >75 years
* Pregnancy
* Epilepsy
* Psychiatric disorders that could possibly influence the study
* Any kind of addiction
* Insufficient knowledge of the language
* Noninvasive ventilation otherwise contraindicated

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Teschler, Dr. med., Principal Investigator — Abteilung Pneumologie - Universitätsklinik, Essen, Germany
Locations (1):
- Abteilung Pneumologie - Universitätsklinik, Ruhrlandklinik, Essen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battisti A, Tassaux D, Bassin D, Jolliet P. Automatic adjustment of noninvasive pressure support with a bilevel home ventilator in patients with acute respiratory failure: a feasibility study. Intensive Care Med. 2007 Apr;33(4):632-8. doi: 10.1007/s00134-007-0550-1. Epub 2007 Feb 24. PMID 17323049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Respiratory insufficiency and hypercapnia requiring noninvasive ventilation. Stable on bi-level CPAP. Both genders. Age >18 and <75years. Requiring EPAP >5cmH2O for upper airway patency, or expected to (e.g. obese patients). Some known to have airway patency at EPAP of 5cmH2O will be included to test for falsely positive response.
Groups:
- AutoVPAP With Addition of AutoEPAP: First AutoVPAP With addition of AutoEPAP then AutoVPAP with EPAP Manually Selected
  Treatment period with conventional device modified to enable algorithm for automatically applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter during a single night of polysomnography following randomisation.
- AutoVPAP With EPAP Manually Selected: "First AutoVPAP With EPAP Manually Selected then AutoVPAP With Addition of AutoEPAP.
  A period of treatment using conventionally applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter during a single night of polysomnography following randomisation.
Period: First Intervention (1 Night)
Arm/Group | AutoVPAP With Addition of AutoEPAP | AutoVPAP With EPAP Manually Selected
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0
Period: Second Intervention(1 Night)
Arm/Group | AutoVPAP With Addition of AutoEPAP | AutoVPAP With EPAP Manually Selected
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Treatment period with conventional device modified to enable algorithm for automatically applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter during a single night of polysomnography following randomisation.
Arm/Group | All Participants
Number analyzed (Participants) | 21
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 19-30 | 2
  Age in years: 31-40 | 0
  Age in years: 41-50 | 1
  Age in years: 51-60 | 7
  Age in years: 61-70 | 7
  Age in years: 71-80 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Region of Enrollment [Number; unit: count of participants]
  Germany | 21
FEV1(%predicted) [Median (Inter-Quartile Range); unit: %predicted] | 37.5 [22 to 59]
FEV1/FVC [Median (Inter-Quartile Range); unit: %] | 52 [44.3 to 56]

OUTCOME MEASURES:

1. Primary Outcome: Index of Apneoas Plus Hypopnoeas Per Hour of Sleep (AHI)
Description: The AHI is a count of the number of pauses during sleep a person experiences. The total number of apneas/ hypopneas (sleep pauses) are divided by the total sleep time to get an index for that night
Time Frame: On completion of each consecutive night of polysomnography.
Measure: Mean (Standard Deviation); unit: Events per hour of sleep
Groups:
- Automatic Algorithm - AutoVPAP With Addition of AutoEPAP: Treatment period with conventional device modified to enable algorithm for automatically applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter during a single night of polysomnography following randomisation.
- Conventional Therapy - AutoVPAP With EPAP Manually Selected: A period of treatment using conventionally applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter during a single night of polysomnography following randomisation.
Arm/Group | Automatic Algorithm - AutoVPAP With Addition of AutoEPAP | Conventional Therapy - AutoVPAP With EPAP Manually Selected
Number analyzed (Participants) | 21 | 21
Events per hour of sleep | 1.3 (2.3) | 1.7 (2.8)

2. Secondary Outcome: Mean SpO2
Description: During sleep, pulse oximetery is recorded through a sensor on the participants finger
Time Frame: On completion of each night of 2 consecutive nights polysomnography.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Automatic Algorithm - AutoVPAP With Addition of AutoEPAP | Conventional Therapy - AutoVPAP With EPAP Manually Selected
Number analyzed (Participants) | 21 | 21
Percent | 92 (3) | 93 (3)

ADVERSE EVENTS:
Time Frame: The intervention took place over 2 nights of polysomnography. No adverse events occurred for any patient on any night polysomnography.
Groups:
- Automatic Algorithm - AutoVPAP With Addition of AutoEPAP: Treatment period with conventional device modified to enable algorithm for automatically applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter
- Conventional Therapy - AutoVPAP With EPAP Manually Selected: A period of treatment using conventionally applied Expiratory Positive Airway Pressure
  AutoVPAP: Implementation of automated algorithm for adjustment of conventional device parameter
Arm/Group | Automatic Algorithm - AutoVPAP With Addition of AutoEPAP | Conventional Therapy - AutoVPAP With EPAP Manually Selected
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

LIMITATIONS AND CAVEATS:
Exclusion of patients whose fundamental disorder was sleep-disordered breathing with an incidental diagnosis of COPD or of OHS and only moderate obesity, and without other supporting evidence, turned out not to be practicable for all cases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No